CLINICAL TRIAL: NCT03956446
Title: Antibiotic Therapy for Patients With Tick-borne Encephalitis and Borrelial Antibodies in Serum
Brief Title: Tick-borne Encephalitis and Borrelial Antibodies in Serum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Principal Investigator, Daša Stupica, Prinicipal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBE-BB prospect
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Tick Borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Doxycycline; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Doxycycline, Doxy® (Active Comparator): Beside symptomatic therapy, patients will receive oral doxycycline 100 mg (Doxy®) twice daily. Patients will answer a questionnaire asking about the presence and frequency of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia.
  Interventions: Drug: Doxycycline; Drug: Symptomatic therapy; Other: Questionnaire
- No antibiotics (Other): Patients will receive symptomatic therapy (paracetamol, Lekadol®, granisetron, Kytril®, metamizol, Analgin®, parenteral hydration with saline). Patients will answer a questionnaire asking about the presence and frequency of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia.
  Interventions: Drug: Symptomatic therapy; Other: Questionnaire
- Healthy controls (Other): Patients will be asked to refer a spouse to serve as a control. If unmarried they will be asked to refer a family member or a friend of +/- 5 years to serve as a control. Control subjects will be asked to answer a questionnaire asking about the presence and frequency of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Drug: Doxycycline — Beside symptomatic therapy, patients will receive oral Doxycycline 100 mg, Doxy® twice daily.
  Arms: Doxycycline, Doxy®
Drug: Symptomatic therapy — Patients will receive symptomatic therapy with antipyretics, analgetics, antiemetics, and parenteral hydration: metamizole, Analgin®, paracetamol, Lekadol®, thiethylperazine, Kytril®, saline. Questionnaire Subjects will be asked to answer a questionnaire asking about the presence and frequency of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia.
  Arms: Doxycycline, Doxy®; No antibiotics
Other: Questionnaire — Subjects will be asked to answer a questionnaire asking about the presence and frequency of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia.

SUMMARY:
In Slovenia, tick-borne encephalitis and Lyme borreliosis are both endemic diseases with high incidence rates and they are both transmitted by a bite of infected Ixodes ricinus tick. In clinical practice, tick-borne encephalitis is confirmed by demonstration of tick-borne encephalitis antibodies in serum of a patient with compatible clinical presentation and cerebrospinal pleocytosis. Patients with Lyme meningitis or meningoradiculitis also have cerebrospinal pleocytosis, however the presence of borrelial antibodies in serum does not attest Lyme neuroborreliosis. Patients with tick-borne encephalitis and positive borrelial antibodies in serum, but not fulfilling criteria for Lyme neuroborreliosis, are often being treated with antibiotics in several European countries due to the possibility of double infection. The investigators hypothesise that such patients do not benefit from antibiotics. Such an approach may appear safe regarding the possibility of borrelial infection, however it can also be associated with detrimental consequences such as antibiotic related adverse reactions, negative epidemiological impact on bacterial resistance, and intravenous catheter related complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* clinical picture compatible with tick-borne encephalitis,
* clear cerebrospinal fluid,
* cerebrospinal pleocytosis (leucocytes in cerebrospinal fluid >5 x 106/)L,
* positive serum immunoglobulin M (IgM) and immunoglobulin G (IgG) antibodies against tick-borne encephalitis virus,
* positive serum IgG antibodies against Lyme borreliae.

Exclusion Criteria:

* isolation of B.burgdorferi sensu lato from cerebrospinal fluid,
* positive intrathecal borrelial antibody production index,
* seroconversion of borrelial IgG antibodies,
* presence of erythema migrans and/or borrelial lymphocytoma in the last month,
* Bannwarth syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with objective manifestations of Lyme borreliosis | one year
  At each visit physical examination will be performed and clinical signs indicating objective manifestations of Lyme borreliosis, such as erythema migrans, will be searched for.
Frequency of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia | one year

CONTACTS AND LOCATIONS:
Overall Officials: Daša Stupica, MD PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia